CLINICAL TRIAL: NCT01770938
Title: Effects of Phototherapy by Low-level Light-emitting Diode Therapy (LEDT) on Clinical, Biochemical, Biomechanical, Histologic and Genetic Responses of Muscle Performance of Young Males Submitted to Physical Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Centro de Pequisas de Ótica e Fotônica (Other)
Responsible Party: Principal Investigator, Cleber Ferraresi, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 0326.0.135.000-11
Record Dates: First submitted 2012-09-15; First posted 2013-01-18 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Light-emitting diode therapy; Muscle performance; Gene expression; Functional performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Effective light-emitting diode therapy and training (Active Comparator): Effects of effective light-emitting diode therapy therapy on muscle performance of young males submitted to physical strength training
  Interventions: Device: Effective light-emitting diode therapy
- Placebo light-emitting diode therapy and training (Placebo Comparator): Effects of placebo light-emitting diode therapy on muscle performance of young males submitted to physical strength training
  Interventions: Device: Placebo light-emitting diode therapy

INTERVENTIONS:
Device: Effective light-emitting diode therapy
  Other Names: LED; LED therapy; Light-emitting diode therapy
  Arms: Effective light-emitting diode therapy and training
Device: Placebo light-emitting diode therapy
  Other Names: LED; LED therapy; Light-emitting diode therapy
  Arms: Placebo light-emitting diode therapy and training

SUMMARY:
Muscle performance is largely influenced by modulations in gene expressions of muscle tissue. In this context, light-emitting diode therapy (LEDT) has been used to improve muscle performance in experimental models and human researches. Thereby, the investigators examined modulations in gene expression of muscle tissue as well as biochemical, biomechanic and histologic adaptations influenced by exercise associated to LEDT.

DETAILED DESCRIPTION:
This study assessed muscle performance in isokinetic dynamometry and led press device, gene expression by RT-PCR, lactate, creatine kinase and morphology of muscle tissue by immunohistochemical analysis

ELIGIBILITY:
Inclusion Criteria:

* healthy males aged between 18 and 28 years with a body mass index (BMI) equal to or less than 26 kg/m2,
* moderated pattern of physical activity

Exclusion Criteria:

* previous injury to the femoral quadriceps or hamstring muscles (within 6 months prior to study),
* osseous or articular disorder in the lower limbs,
* cardiovascular system disorders,
* systemic disease, and
* taking prescription medicines or using dietary supplements such as muscle mass builders.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Modulations on muscle gene expression by RT-PCR | 12 weeks

SECONDARY OUTCOMES:
Muscle performance in leg press device | 12 weeks
Muscle performance in leg extension device | 12 weeks
Muscle performance in isokinetic dynamometer | 12 weeks
Gene expression | 12 weeks
  Gene expression of muscle tissue by RT-PCR

OTHER OUTCOMES:
Immunohistochemical analysis | 12 weeks
  Immunohistochemical analysis to quantify morphology and cells of muscle tissue as satellite cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cleber Ferraresi, MSc, Principal Investigator — Universidade Federal de Sao Carlos; Nivaldo A Parizotto, PhD, Study Director — Universidade Federal de Sao Carlos; Vanderlei S Bagnato, PhD, Study Director — University of Sao Paulo
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010